CLINICAL TRIAL: NCT04220541
Title: Investigation of the Effects of Different Exercise Programs on Patients With Chiari Malformation Type 1
Brief Title: Investigation of the Effects of Exercise on Patients With Chiari Malformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19155
Record Dates: First submitted 2020-01-04; First posted 2020-01-07 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Chiari Malformation Type I; Proprioceptive Disorders; Coordination and Balance Disturbances; Syringomyelia; Basilar Invagination; Exercise Addiction; Atlanto-Axial Subluxation
MeSH Terms: conditions — Arnold-Chiari Malformation; Somatosensory Disorders; Syringomyelia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor learning based exercise group (Experimental)
  Interventions: Behavioral: Motor learning based exercise
- Symptomatic exercise group (Experimental)
  Interventions: Behavioral: Motor learning based exercise

INTERVENTIONS:
Behavioral: Motor learning based exercise — Symptomatic exercise

SUMMARY:
Chiari Malformation (CM) is a posterior brain anomaly caused by the displacement of the brain stem and cerebellum into the cervical spinal canal. There are 8 types of Chiari malformations described today that vary according to the severity of the anomaly.

In CM Type 1, cerebrospinal fluid (CSF) circulation deteriorated along with the foramen magnum and the cerebellar tonsillar decreased to at least 5 mm below the foramen magnum. Depending on this situation, headache, cerebellar findings, muscle strength, and sensory loss and so on. and adversely affect the daily life of the patient.

When establishing an exercise program for the symptoms of CM type 1, it should be taken into consideration that somatosensory, visual, vestibular system and cerebellum are in close relationship with each other and balance and coordination result from this close relationship.

When the literature is reviewed for exercise programs aimed at reducing instability in the cervical region, it is seen that 80% of the stability of the cervical spine originates from the muscular system and its importance in the treatment process is being investigated more and more day by day. However, no randomized controlled study was performed on these subjects. This study was planned to investigate the effects of two different exercise programs on pain, balance, coordination, proprioception, functional capacity, body posture, daily life activities and quality of life. The study was planned to involve at least 20 individuals with CM Type 1 who were not surgical indications in the 18-65 age range. The study was designed as a randomized, self-controlled study. Demographic data and characteristics of the subjects who meet the inclusion criteria and agree to participate in the study will be recorded at the beginning of the study. Patients will be evaluated in two different time periods. The first evaluations will be performed on the first day when patients are referred to rehabilitation by the physician. Following this assessment, all patients will be assigned numbers, which will be divided into two groups using a simple randomization method in the form of drawing lots. A total of 18 sessions 3 times a week for six weeks, the first group will receive symptomatic exercise program and the second group will focus on the deep muscles in the cervical region, especially the stabilizer, and a "Motor learning-based" exercise program that includes gradual control of these muscles. After 6 weeks, the first evaluations will be repeated in both groups.

ELIGIBILITY:
Inclusion Criteria:

* The study was planned to involve at least 20 individuals with CM Type 1 who were not surgical indications in the 18-65 age range.

Exclusion Criteria:

* Motor type defect due to CM Type 1,
* Presence of primary neurological disease other than CM Type 1, severe cognitive impairment (> 24 from the Mini Mental State Assessment),
* peripheral vestibular problem and history of orthopedic surgery,
* patients who had musculoskeletal problems in the last 6 months and who received physiotherapy rehabilitation program in the last 6 months,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 weeks
  The Neck Disability Index (NDI) is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. ... Questions include activities of daily living, such as: personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration and headache.
Visual Analog Scale | 1 week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.

SECONDARY OUTCOMES:
Berg Balance Scale | 6 weeks
  The BBS is a qualitative measure that assesses balance via performing functional activities such as reaching, bending, transferring, and standing that incorporates most components of postural control: sitting and transferring safely between chairs; standing with feet apart, feet together, in single-leg stance, and feet in the tandem Romberg position with eyes open or closed; reaching and stooping down to pick something off the floor. Each item is scored along a 5-point scale, ranging from 0 to 4, each grade with well-established criteria. Zero indicates the lowest level of function and 4 the highest level of function. The total score ranges from 0 to 56.
Posture Screen Mobile | 24 hours
  PostureScreen Mobile allows you to accurately assess and analyze posture in seconds. Report provides front and side view photos clearly describing postural faults.
Short Form-36 | 4 weeks
  As part of the Medical Outcomes Study (MOS), a multi-year, multi-site study to explain variations in patient outcomes, RAND developed the 36-Item Short Form Health Survey (SF-36). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.
International Cooperative Ataxia Rating Scale | 6 weeks
  The International Cooperative Ataxia Rating Scale (ICARS) is an outcome measure that was created in 1997 by the Committee of the World Federation of Neurology with the goal of standardizing the quantification of impairment due to cerebellar ataxia. The scale is scored out of 100 with 19 items and 4 subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Higher scores indicate higher levels of impairment.
  Intended Population

CONTACTS AND LOCATIONS:
Locations (1):
- Ceyhun Türkmen, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No